CLINICAL TRIAL: NCT06150482
Title: Healthcare Utilization in Liver Cirrhosis Patients, a Multicenter Retrospective Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Gelre Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-2857-A-2
Record Dates: First submitted 2023-05-23; First posted 2023-11-29 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2024-12

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Multicenter, retrospective cohort study investigating healthcare utilization in compensated and decompensated liver cirrhosis patients, including disease course and characteristics associated with healthcare utilization and, for example psychosocial factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* Liver cirrhosis, based on biopsy, fibroscan or diagnostic imaging data

Exclusion Criteria:

* Known malignancy with hepatic metastasis at baseline
* Liver transplantation at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of liver cirrhosis related outpatient contacts before liver cirrhosis complications | 2 years before complication, death or loss to follow-up
Number of liver cirrhosis related radiographic imaging before liver cirrhosis complications | 2 years before complication, death or loss to follow-up
Number of liver cirrhosis related esophagogastroscopies before liver cirrhosis complications | 2 years before complication, death or loss to follow-up
Number of liver cirrhosis related elastographies before liver cirrhosis complications | 2 years before complication, death or loss to follow-up

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Gelre Ziekenhuizen, Apeldoorn, Gelderland
  - Maastricht University Medical Center, Maastricht, Limburg

IPD SHARING:
Plan to Share IPD: Undecided